CLINICAL TRIAL: NCT00110682
Title: A Randomized, Parallel-Group, Vehicle-Controlled, Double-Blind Study of Topical Imiquimod 5% Cream Used as an Adjunct to Cryotherapy in the Management of Actinic Keratoses, With a Long-Term (1 Year) Follow-Up
Brief Title: Study of Imiquimod 5% Cream in Addition to Cryotherapy in the Management of Actinic Keratoses
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Derm Research @ 888 Inc. (Industry)
Collaborators: 3M (Industry)
Responsible Party: D Richard Thomas, Department of Dermatology and Skin Science
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DR 2004-05
Record Dates: First submitted 2005-05-12; First posted 2005-05-13 (Estimated); Last update posted 2008-04-24 (Estimated); Status verified 2008-04

CONDITIONS: Keratosis; Actinic Keratosis
Keywords: Actinic Keratosis; Cryotherapy; Imiquimod
MeSH Terms: conditions — Keratosis; Keratosis, Actinic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Imiquimod used as an adjunct to cryotherapy

SUMMARY:
Study Aims:

* To compare the long-term efficacy and safety of imiquimod versus vehicle used as an adjunct to cryotherapy.
* To assess and compare the recurrence rate and time to recurrence of the 2 different treatment groups.

Hypothesis: The imiquimod arm will produce a more prolonged clearing of Actinic Keratoses (AK) compared to the vehicle arm.

DETAILED DESCRIPTION:
Evaluation of: (i) topical imiquimod 5% cream or (ii) vehicle cream used two times weekly for eight weeks starting two weeks post cryotherapy.

Study Aims:

* To assess and compare the recurrence rate and time to recurrence of the 2 different treatment groups.
* To assess and compare the efficacy of the 2 different treatment groups.
* To assess and compare the safety of the 2 different treatment groups.

Study Design: 6 visits over 62 weeks

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of actinic keratosis with 4 or more discreet lesions on the face or balding scalp. Lesions must be within a treatment area not exceeding 50 cm2 (combined total must not exceed 50 cm2)
* Women of childbearing potential using appropriate contraceptive methods

Exclusion Criteria:

* Previous treatments with imiquimod for AK in the prescribed area within the past 5 months or cryosurgery in the same area within the past 4 weeks.
* Patients unwilling to stay out of the sun or wear protective clothing or to use sunscreen with a minimum of SPF 15 during the study.
* Basal or squamous cell carcinomas in the prescribed treatment area in the past 2 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-04; Primary Completion 2006-10 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Recurrence rate and time to recurrence of lesions

SECONDARY OUTCOMES:
Time to reach treatment success
Percentage of patients who clear
Patient improvement assessment

CONTACTS AND LOCATIONS:
Overall Officials: Yves Poulin, MD FRCPC, Principal Investigator — Centre de Recherche Dermatologique du Quebec Metropolitaine; Jerry KL Tan, MD FDRPC, Principal Investigator — U. of Western Ontario, Windsor Ontario; Richard Thomas, MD FRCPC, Principal Investigator — Derm Research @ 888 Inc.
Locations (3):
- Canada (3):
  - DermResearch @ 888 Inc, Vancouver, British Columbia
  - Windsor Clinical Research, Windsor, Ontario
  - Centre de Recherche Dermatologique, CRDQ, Sainte-Foy, Quebec